CLINICAL TRIAL: NCT02259920
Title: Open Label, Randomized, Single-dose, Five-way Crossover Study to Investigate the Regional Drug Absorption of 80 mg KUC-7483 CL Administered Via an Enterion™ Capsule Compared to an Immediate Release Formulation in Healthy Male Volunteers.
Brief Title: Study to Investigate the Regional Drug Absorption of KUC-7483 CL Administered Via an Enterion™ Capsule Compared to an Immediate Release Formulation in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1207.2
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (5):
- Treatment A (Active Comparator): KUC 4783 CL, immediate release tablets
  Interventions: Drug: KUC 7483 CL, immediate release tablet
- Treatment B (Experimental): KUC 4783 CL delivered as a particulate formulation to the distal small bowel
  Interventions: Drug: KUC 7483 CL, particulate formulation; Device: Enterion™ capsule
- Treatment C (Experimental): KUC 4783 CL delivered as a particulate formulation to the ascending colon
  Interventions: Drug: KUC 7483 CL, particulate formulation; Device: Enterion™ capsule
- Treatment D (Experimental): KUC 4783 CL delivered as a solution formulation to the ascending colon
  Interventions: Drug: KUC 7483 CL, solution formulation; Device: Enterion™ capsule
- Treatment E (Experimental): KUC 4783 CL delivered as a solution formulation to the descending colon
  Interventions: Drug: KUC 7483 CL, solution formulation; Device: Enterion™ capsule

INTERVENTIONS:
Drug: KUC 7483 CL, immediate release tablet
  Arms: Treatment A
Drug: KUC 7483 CL, particulate formulation
  Arms: Treatment B; Treatment C
Drug: KUC 7483 CL, solution formulation
  Arms: Treatment D; Treatment E
Device: Enterion™ capsule
  Arms: Treatment B; Treatment C; Treatment D; Treatment E

SUMMARY:
Study to determine and compare the absorption of KUC 7483 CL from different regions of the GI tract with the immediate release formulation and to compare the absorption of particulate versus solution formulations from the ascending colon

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males, according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG, clinical laboratory tests
   * No clinically significant findings
   * No evidence of a clinically relevant concomitant disease
2. Age ≥18 and ≤65 years
3. BMI ≥18.5 and ≤29.9 kg/m2
4. Subjects must be able to demonstrate the ability to swallow an empty size 000 gelatin capsule
5. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. History of gastrointestinal surgery, with the exception of Appendicectomy unless it was performed within the previous 12 months
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) to any drug including the study drug (KUC-7483 CL) and similar drugs which is deemed relevant to the trial as judged by the investigator
7. Use of prescription or non-prescription drugs (including vitamins and natural herbal remedies e.g. St Johns Wort) from 14 days prior to the start of the study until the end of the final study period. Occasional use of paracetamol (up to 4g per day) is permitted throughout the study
8. Participation in another trial with an investigational drug within four months prior to administration or during the trial
9. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day). A breath carbon monoxide reading of greater than 20ppm
10. Inability to refrain from smoking on trial days
11. Regular alcohol consumption >21 units per week units per week (1 Unit = ½ pint beer, a 25ml shot of 40% spirit or a 125ml glass of wine)
12. Subjects who have ever sought advice from a physician or counselor for abuse or misuse of alcohol, non-medicinal drugs or other substances of abuse e.g. solvents
13. Any current or previous use of Class A drugs such as opiates, cocaine, ecstasy, lysergic acid diethylamide, and amphetamines (Class B).

    Volunteers who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs of abuse test and have been abstinent for at least 12 months
14. Positive drugs of abuse result
15. Blood donation (more than 100 mL within three months prior to administration or during the trial)
16. Excessive physical activities outside a subjects normal routine (within one week prior to administration or during the trial until after the post-study medical)
17. Unable to eat all elements of a standard meal
18. Any laboratory value outside the reference range of clinical relevance as determined by the Investigator
19. Radiation exposure from clinical trials, including that from the present study and from diagnostic X-rays but excluding background radiation, exceeding 5mSv in the last twelve months or 10mSv in the last five years. No subject whose occupational exposure is monitored will participate in the study
20. Acute diarrhea, or constipation in the 14 days before the predicted first study day. If screening occurs >14 days before first study day, this criterion is to be determined on first study day. Diarrhea will be defined as the passage of liquid faeces and/or a stool frequency of greater than three times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day
21. Presence of non-removable metal objects such as metal plates, screws etc. in abdominal region of the body
22. Subjects will be excluded from the study if they are considered by the investigator to be at risk of transmitting through blood and other body fluids the agents responsible for AIDS (Acquired Immunodeficiency Syndrome) or other sexually transmitted disease or hepatitis. This will be achieved by the use of a card (similar to that used by the National Blood Transfusion Service) which asks a potential subject if they have reason to believe that they may fall into any category included on the card. If the verbal answer is in the affirmative then they will be excluded from the study
23. Positive hepatitis B virus, hepatitis C virus or HIV results

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-12; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
Cmax(maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 24 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 24 hours after drug administration
λz (terminal rate constant of the analyte constant in plasma) | up to 24 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 24 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 24 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 24 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 24 hours after drug administration
Aet1-t2 (amount of the analyte that is eliminated in urine from the time point t1 until time point t2) | up to 24 hours after drug administration
fet1-t2 (fraction of administered drug excreted unchanged in urine from the time point t1 until time point t2) | up to 24 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte determined from the time point t1 until time point t2) | up to 24 hours after drug administration
Number of subjects with adverse events | up to 8 days after last drug administration